CLINICAL TRIAL: NCT06919302
Title: An Innovative Technology-based Approach to Translating Clinical Practice Guidelines of Nutrition Therapy in Primary Care: The Coronary Heart Effectiveness Assessment of the Portfolio Diet in Primary Care (CHEAP) Trial
Brief Title: The Effect of a Digital Heart Health App and Lifestyle Intervention for Heart Disease in Primary Care.
Acronym: CHEAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Laura Chiavaroli, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB-44995
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factors; Dyslipidemia; Cholesterol; Major Cardiovascular Event
Keywords: randomized controlled trial; digital heart health program; heart health app; web-based app; large-scale study
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to the nature of the treatment when analyzing data (i.e., will not know the treatment assignment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Digital Heart Health Program + Standard of Care (Experimental)
  Interventions: Behavioral: Digital Heart Health Program

INTERVENTIONS:
Behavioral: Digital Heart Health Program — The digital heart health program will include the web-based app, which will deliver the intervention through interactive features (dashboard, goal setting, gamification, nudges, etc.) and will be supported by a 16-session synchronous online behaviour change program and provision of key study foods.
  Arms: Digital Heart Health Program + Standard of Care

SUMMARY:
Despite the availability of medications, many people around the world continue to live with long-term health problems like heart disease, stroke and diabetes. In Canada, heart disease is a leading cause of death. Managing these health issues can be done by changing diet and lifestyle. Specific ways of eating have been proven to improve risk for heart disease and stroke. However, because doctors often have limited time, nutrition education, and lack of tools for counseling patients on nutrition, they can often only provide minimal support to help patients make necessary lifestyle changes. Digital tools and mobile applications offer an opportunity to involve doctors and patients in delivering nutrition interventions. This approach has the potential to save time, provide education, and reduce healthcare costs. This study is being done to understand the effect of a digital heart health program added to standard of care, compared with standard of care alone on heart health. All eligible participants in this study will be randomized (determined by chance) to one of two possible interventions: 1) a digital heart health program + standard of care; 2) standard of care. Standard is care is defined as the best practice based on guidelines for the treatment of a condition. All participants will be followed for seven years and will be asked to complete online questionnaires and complete blood work at their nearest LifeLabs clinic, as well as wear a continuous glucose monitor and wrist actigraph (at 3 time points in the first year). In addition, participants randomized to the digital heart health program + standard of care will be expected to use the heart health app and join 16 online synchronous sessions over the first year.

After seven years, the intervention phase of the study will end and the study will become a cohort study. All participants at the 7-year time point will be invited to use the heart health app. As part of the cohort study, participants will be asked to continue completing the same questionnaires online and completing bloodwork at their nearest LifeLabs every four years for the duration of their participation in the cohort study.

The main questions this study aims to answer are:

1. Will a digital heart health program added to standard of care result in a clinically meaningful reduction in blood cholesterol and other risk factors after 1-year compared to standard of care alone?
2. Will a digital heart health program added to standard of care result in a reduction in major cardiovascular events after 7-years compared to standard of care alone?
3. Are the observed effects sustained beyond the 7-years of the intervention?

We hypothesize that the digital heart health program added to standard of care will result in a clinically meaningful reduction in blood cholesterol and other risk factors for heart disease after 1-year and reduce major cardiovascular events after 7-years compared to standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Be taking statin medication with or without other antihyperlipidemic therapy (stable dose for at least 3-months).
* Fall under either of the 2 categories:

  1) Secondary prevention participants: males and females ≥45 years of age with established atherosclerotic cardiovascular disease (ASCVD) defined as at least one of the following: i. Prior myocardial infarction (MI); ii. Acute coronary syndrome (ACS); iii. Stroke/TIA; iv. Coronary revascularization; v. Documented carotid disease (endarterectomy, carotid stenosis ≥50%); vi. Stable angina; vii. Coronary artery disease (CAD) by angiography; viii. Peripheral artery disease (PAD); ix. Abdominal aortic aneurysm (AAA)

  2) High-risk primary prevention participants: males and females ≥50 years of age plus type 2 diabetes requiring treatment with medication and at least one additional risk factor: i. Males ≥55 years of age and females ≥65 years of age; ii. Cigarette smoker or stopped smoking within 3 months before Visit 1; iii. Hypertension and on antihypertensive medication for at least 6-months; iv. Chronic kidney disease (CKD); v. Retinopathy, defined as any of the following: non-proliferative retinopathy, pre-proliferative retinopathy, proliferative retinopathy, maculopathy, advanced diabetic eye disease or a history of photocoagulation
* Be on a stable dose for at least 3-months of all antihyperlipidemic, antihyperglycemic, antihypertensive, and antiobesity therapies.
* Have a family physician in Ontario and a valid Ontario Health Card.
* Have regular access to an online portal
* Be proficient in English.

Exclusion Criteria:

* Major disease expected to result in death within 2 years (except cardiovascular disease)
* Active sever liver disease
* Malabsorption disorders
* Drug or alcohol abuse disorders (within past 6 months)
* Intolerance or allergies to soy protein and tree nuts, peanuts, or seeds
* Planned coronary intervention or any major surgical procedure
* Participation in another clinical trial (within past 3 months)
* End stage renal disease (requirement for peritoneal dialysis or hemodialysis for renal insufficiency or eGFR <30 mL/min)
* Any condition or therapy which might pose a risk to the patient or make participation in the study not be in the best interest of the patient as assessed by the investigator
* Documented severe (New York Heart Association [NYHA] class IV) heart failure
* Mental/psychological impairment expected to affect adherence to the study protocol
* Known AIDS (HIV-positive patients without AIDS are allowed)
* Women planning on becoming pregnant within the first year of the intervention
* Unable to provide informed consent: Appear unable to comprehend the study protocol during the interview process or to understand and communicate in English sufficiently for informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2034-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion achieving a ≥8% reduction in LDL-C or non-HDL-C | from enrollment to 1-year
  Proportion of participants who achieve a ≥8% reduction in LDL-C or non-HDL-C in the intervention group compared to standard of care at 1-year.
  (If this is not achieved, we will then assess the difference in the proportion achieving ≥8% reduction in LDL-C or non-HDL-C and ≥5mmHg reduction in systolic blood pressure. If this is not achieved, we will then assess the difference in the proportion achieving ≥8% reduction in LDL-C or non-HDL-C and ≥10% reduction in the inflammatory marker, CRP.)
Major Cardiovascular Events | from enrollment to 7-years
  Major cardiovascular events in the intervention group compared to standard of care at 7-years.

SECONDARY OUTCOMES:
Dietary Adherence | from enrollment to 1-year and 7-years
  Proportion of participants who achieves ≥12/25-pt Diet Score, in the intervention group compared to standard of care at 1-year and 7-years. The Diet Score will be assessed using the Harvard Willett food frequency questionnaire.
Proportion achieving a ≥8% reduction in LDL-C or non-HDL-C | from enrollment to 7-years
  Proportion of participants who achieve a ≥8% reduction in LDL-C or non-HDL-C in the intervention group compared to standard of care at 7-years.
Proportion achieving established lipid targets for LDL-C or non-HDL-C | from enrollment to 1-year and 7-years
  Proportion of participants who achieve Canadian Cardiovascular Society targets for LDL-C (<2.0mmol/L for primary <1.8mmol/L for secondary prevention) or non-HDL-C (<2.6mmol/L for primary and <2.4mmol/L for secondary prevention) in the intervention group compared to standard of care at 1-year and 7-years.
Blood Lipids | from enrollment to 1-year and 7-years
  Changes in LDL-C, non-HDL-C, HDL-C, triglycerides and apoB levels in the intervention group compared to standard of care at 1-year and 7-years
Changes in Lipid-Lowering Medications | from enrollment to 1-year and 7-years
  Changes in lipid-lowering medications in the intervention group compared to standard of care at 1-year and 7-years
Changes in Glycemia | from enrollment to 1-year and 7-years
  Changes in HbA1c in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Glycemia | from enrollment to 1-year and 7-years
  Changes in fasting blood glucose levels in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Insulin Resistance | from enrollment to 1-year and 7-years
  Changes in HOMA-IR in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Insulin | from enrollment to 1-year and 7-years
  Changes in fasting blood insulin levels in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Measures of Adiposity | from enrollment to 1-year and 7-years
  Changes in body weight in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Measures of Adiposity | from enrollment to 1-year and 7-years
  Changes in body mass index in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Measures of Adiposity | from enrollment to 1-year and 7-years
  Changes in waist circumference in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Systolic Blood Pressure | from enrollment to 1-year and 7-years
  Changes in systolic blood pressure in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Diastolic Blood Pressure | from enrollment to 1-year and 7-years
  Changes in diastolic blood pressure in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Inflammation | from enrollment to 1-year and 7-years
  Changes in c-reactive protein (CRP) levels in the intervention group compared to the standard of care at 1-year and 7-years
Cost-Effectiveness - quality-adjusted life years (QALYs) | from enrollment to 1-year and 7-years
  Changes in quality-adjusted life years (QALYs) assessed using the EQ5D-5L in the intervention group compared to standard of care at 1-year and 7-years
Cost-Effectiveness - medical resource utilization | from enrollment to 1-year and 7-years
  Changes in medical resources utilization (Canadian dollars) in the intervention compared to standard of care at 1-year and 7-years.
  Medical resource utilization encompassing primary care, hospital care, specialist care, and medications for individuals covered by public drug insurance will be obtained from Ontario health administrative databases housed at ICES (formerly the Institute for Clinical Evaluative Sciences).
Cost-Effectiveness - out-of-pocket food and medical costs | from enrollment to 1-year and 7-years
  Changes in out-of-pocket food and medical costs in the intervention group compared to the standard of care at 1-year and 7-years
Cost-utility | from enrollment to 1-year and 7-years
  Costs / point change in QALY in the intervention group compared to the standard of care at 1-year and 7-years

OTHER OUTCOMES:
Changes in Anti-Hypertension Medications | from enrollment to 1-year and 7-years
  Changes in anti-hypertension medications in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Anti-Hyperglycemic Medications | from enrollment to 1-year and 7-years
  Changes in anti-hyperglycemic medications in the intervention group compared to the standard of care at 1-year and 7-years
Changes in Glycaemia | from enrollment to 1-year
  Changes in ambulatory glucose measured via a continuous glucose monitor in the intervention group compared to the standard of care at 1-year
Changes in Sleep | from enrollment to 1-year
  Changes in sleep using actigraphy in the intervention group compared to the standard of care at 1-year
Changes in Sleep | from enrollment to 1-year and 7-years
  Changes in sleep using questionnaires in the intervention group compared to the standard of care at 1-year and 7-years
Safety - Self-Reported Adverse Events | from enrollment to 1-year and 7-years
  Adverse events participants experience in the intervention group compared to the standard of care at 1-year and 7-years
Incidence of Type 2 Diabetes | from enrollment to 7-years
  Incidence of type 2 diabetes in the intervention group compared to the standard of care at 7-years
Type 2 Diabetes Remission | from enrollment to 7-years
  Type 2 diabetes remission in the intervention group compared to the standard of care at 7-years
Incidence of Metabolic Syndrome | from enrollment to 7-years
  Incidence of metabolic syndrome in the intervention group compared to the standard of care at 7-years
Metabolic Syndrome Remission | from enrollment to 7-years
  Metabolic syndrome remission in the intervention group compared to the standard of care at 7-years
Incidence of Hypertension | from enrollment to 7-years
  Incidence of hypertension in the intervention group compared to the standard of care at 7-years
Incidence of Cancer | from enrollment to 7-years
  Incidence of cancer in the intervention group compared to the standard of care at 7-years
Incidence of Dementia | from enrollment to 7-years
  Incidence of dementia in the intervention group compared to the standard of care at 7-years

CONTACTS AND LOCATIONS:
Locations (1):
- C. David Naylor Building, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All outcomes listed will be shared in an anonymous/de-identified format.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available after the anticipated study completion date from 2035 and will remain for 30 years.
Access Criteria: IPD data will be accessible though the University of Toronto Dataverse (https://borealisdata.ca/dataverse/toronto). The metadata record of our dataset will be public, however access to the data will be restricted. Users will need to request access using the contact information provided in order to view and download our restricted files.